CLINICAL TRIAL: NCT00983229
Title: Position of Supraglottic Airway as a Conduit for Tracheal Intubation - A Comparison of CTrach, Intubating LMA and I-gel Supraglottic Airway
Brief Title: Comparison of CTrach, Intubating Laryngeal Mask Airway (ILMA) and I-gel for Tracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Health and Social Care Trust (Other Government)
Responsible Party: Pavel Michalek, MD PhD DESA, Consultant Anaesthetist, Northern Health and Social Care Trust, Antrim Area Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09/NIR03/44
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-10

CONDITIONS: Intubation
Keywords: difficult airway; fibreoptic intubation; supraglottic airways; laryngeal mask airway
MeSH Terms: interventions — Intubation, Intratracheal; Intubation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CTrach (Active Comparator): 1. Induction to GA with 1mcg/kg fentanyl, and 1-3 mg/kg of propofol to loss of verbal contact and neuromuscular relaxation with 0.5 mg/kg of atracurium.
  2. Direct laryngoscopy, evaluation of laryngeal view grade according to Cormack-Lehane classification.
  3. Insertion of CTrach (sizes 3,4 or 5), establishment of ventilation.
  4. Direct evaluation of laryngeal view through CTrach
  5. Tracheal intubation through CTrach LMA
  6. Maintenance of anaesthesia with 02, air and sevoflurane 1-2 MAC and positive pressure ventilation
  7. At the end of surgery patient will be awoken as normal. Any sign of trauma to the oral cavity and airways and gastric fluid in trachea will be noted.
  Interventions: Procedure: Tracheal intubation
- Intubating Laryngeal Mask Airway (ILMA) (Active Comparator): 1. Induction to GA with 1mcg/kg fentanyl, and 1-3 mg/kg of propofol to loss of verbal contact and neuromuscular relaxation with 0.5 mg/kg of atracurium.
  2. Direct laryngoscopy, evaluation of laryngeal view grade according to Cormack-Lehane classification.
  3. Insertion of ILMA (sizes 3,4 or 5), establishment of ventilation.
  4. Evaluation of laryngeal view through ILMA using fibrescope
  5. Tracheal intubation through ILMA using fibrescope.
  6. Maintenance of anaesthesia with 02, air and sevoflurane 1-2 MAC and positive pressure ventilation
  7. At the end of surgery patient will be awoken as normal. Any sign of trauma to the oral cavity and airways and gastric fluid in trachea will be noted.
  Interventions: Procedure: Tracheal intubation
- I-gel (Active Comparator): 1. Induction to GA with 1mcg/kg fentanyl, and 1-3 mg/kg of propofol to loss of verbal contact and neuromuscular relaxation with 0.5 mg/kg of atracurium.
  2. Direct laryngoscopy, evaluation of laryngeal view grade according to Cormack-Lehane classification.
  3. Insertion of I-gel (sizes 3,4 or 5), establishment of ventilation.
  4. Evaluation of laryngeal view through I-gel using fibrescope
  5. Tracheal intubation through I-gel using fibrescope
  6. Maintenance of anaesthesia with 02, air and sevoflurane 1-2 MAC and positive pressure ventilation
  7. At the end of surgery patient will be awoken as normal. Any sign of trauma to the oral cavity and airways and gastric fluid in trachea will be noted.
  Interventions: Procedure: Tracheal intubation

INTERVENTIONS:
Procedure: Tracheal intubation — Insertion of a plastic tube under direct vision (built-in camera, intubating fibrescope) into trachea.
  Other Names: intubation; insertion of tracheal tube

SUMMARY:
Various supraglottic airways may be used as a dedicated airway for insertion of intubating fibrescope and tracheal intubation in the patients with difficult to manage airways (Difficult Airway Society Guidelines).

The investigators aim to compare three different types of supraglottic device as a conduit for tracheal intubation - CTrach optical laryngeal mask, Intubating laryngeal mask airway and I-gel supraglottic airway. Null hypothesis for this study is that all three devices will perform without statistical difference in the means of success rate and time needed for their insertion and tracheal intubation.

DETAILED DESCRIPTION:
Supraglottic airway devices such as I-LMa, Igel and LMA Ctrach are designed to create a "dedicated" airway which safely allows both spontaneous and controlled ventilation. The use of supraglottic airways can allow planned fibreoptic intubations in expected difficult cases and can provide an emergency airway in cases of unexpected difficult airway.

The ILMA (Intavent Orthofix Ltd.,Wokingham, UK) has been designed for either blind or fibrescope-guided tracheal intubation, in patients with expected and unexpected difficult airway. Since its development in 1997, it has been used for both blind and fibrescope-guided tracheal intubations in the patients with difficult airway. The ILMA is currently a 'gold standard' in supraglottic airways used for tracheal intubation.

The I-gel (Intersurgical Ltd., Wokingham, UK) is a newer dedicated airway device, which with its wide bore allows direct passage of a tracheal tube.

The CTrach (The Laryngeal Mask Company,Singapore) is a newer device for airway management. It has special optical fibres built-in inside its bowl and a liquid crystal display which allows views of the larynx while the endotracheal tube is being placed.

With reference to these supraglottic airway devices, only a small number of case reports detail tracheal intubation through an I-gel in patients with difficult airways. There have been manikin studies comparing ILMA and CTrach, and some descriptive studies on the use of CTrach in patients with predicted difficult airways- but no studies comparing the performance of these devices in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients
* Age 18-89 years, males and females
* Elective surgical patients needing tracheal intubation

Exclusion Criteria:

* ASA IV or V patients
* Emergency surgical procedures
* Patients at increased risk of aspiration

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Success rate of tracheal intubation (%) | After successful insertion of tracheal tube

SECONDARY OUTCOMES:
Time needed for successful insertion of a supraglottic device | After insertion
Total time needed for successful tracheal intubation through a device | After insertion
Fibreoptic view following to supraglottic device insertion | After insertion of SGA
Complication rate - sore throat, difficulty swallowing, hoarseness, numb tongue, nausea | at 1 h after operation, at 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Michalek, MD,PhD,DESA, Principal Investigator — Northern HSC Trust
Locations (1):
- Antrim Area Hospital, Antrim, Antrim, United Kingdom

REFERENCES:
- [Background] Campbell J, Michalek P, Deighan M. I-gel supraglottic airway for rescue airway management and as a conduit for tracheal intubation in a patient with acute respiratory failure. Resuscitation. 2009 Aug;80(8):963. doi: 10.1016/j.resuscitation.2009.04.037. Epub 2009 Jun 10. No abstract available. PMID 19520483
- [Background] Michalek P, Hodgkinson P, Donaldson W. Fiberoptic intubation through an I-gel supraglottic airway in two patients with predicted difficult airway and intellectual disability. Anesth Analg. 2008 May;106(5):1501-4, table of contents. doi: 10.1213/ane.0b013e31816f22f6. PMID 18420867
- [Background] Sreevathsa S, Nathan PL, John B, Danha RF, Mendonca C. Comparison of fibreoptic-guided intubation through ILMA versus intubation through LMA-CTrach. Anaesthesia. 2008 Jul;63(7):734-7. doi: 10.1111/j.1365-2044.2008.05481.x. PMID 18582259
- [Background] Ferson DZ, Rosenblatt WH, Johansen MJ, Osborn I, Ovassapian A. Use of the intubating LMA-Fastrach in 254 patients with difficult-to-manage airways. Anesthesiology. 2001 Nov;95(5):1175-81. doi: 10.1097/00000542-200111000-00022. PMID 11684987
- [Background] Charters P, O'Sullivan E. The 'dedicated airway': a review of the concept and an update of current practice. Anaesthesia. 1999 Aug;54(8):778-86. doi: 10.1046/j.1365-2044.1999.00888.x. PMID 10460531
- [Background] Pandit JJ, MacLachlan K, Dravid RM, Popat MT. Comparison of times to achieve tracheal intubation with three techniques using the laryngeal or intubating laryngeal mask airway. Anaesthesia. 2002 Feb;57(2):128-32. doi: 10.1046/j.0003-2409.2001.02401.x. PMID 11871949
- [Background] Joo HS, Kapoor S, Rose DK, Naik VN. The intubating laryngeal mask airway after induction of general anesthesia versus awake fiberoptic intubation in patients with difficult airways. Anesth Analg. 2001 May;92(5):1342-6. doi: 10.1097/00000539-200105000-00050. PMID 11323374
- [Background] Ng BS, Goy RW, Bain JA, Chen FG, Liu EH. The impact of manual in-line stabilisation on ventilation and visualisation of the glottis with the LMA CTrach: a randomised crossover trial. Anaesthesia. 2009 Aug;64(8):894-8. doi: 10.1111/j.1365-2044.2009.05935.x. PMID 19604194
- [Background] Liu EH, Goy RW, Lim Y, Chen FG. Success of tracheal intubation with intubating laryngeal mask airways: a randomized trial of the LMA Fastrach and LMA CTrach. Anesthesiology. 2008 Apr;108(4):621-6. doi: 10.1097/ALN.0b013e318167af61. PMID 18362593
- [Background] Liu EH, Goy RW, Chen FG. An evaluation of poor LMA CTrach views with a fibreoptic laryngoscope and the effectiveness of corrective measures. Br J Anaesth. 2006 Dec;97(6):878-82. doi: 10.1093/bja/ael252. Epub 2006 Sep 19. PMID 16984953